CLINICAL TRIAL: NCT02770261
Title: A Multi-center, Randomized, Double-blind, Parellel Phase III Clinical Trial to Evaluate the Efficacy and Safety of DP-R208 and Each Monotherapy in Patients With Hypertension and Primary Hypercholesterolemia.
Brief Title: Phase III Clinical Trial to Evaluate the Efficacy and Safety of DP-R208 and Each Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DP-CTR208-III-03
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Hypertension; Cholesterolemia
Keywords: DP-R208
MeSH Terms: conditions — Hypertension | interventions — candesartan; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CR group (Experimental): DP-R208+Candesartan 32mg pla+Rosuvastatin 20mg pla
  Interventions: Drug: DP-R208; Drug: Candesartan32mg Placebo; Drug: Rosuvastatin 20mg Placebo
- CP group (Active Comparator): DP-R208 pla+Candesartan 32mg+Rosuvastatin 20mg pla
  Interventions: Drug: Candesartan32mg; Drug: DP-R208 Placebo; Drug: Rosuvastatin 20mg Placebo
- PR group (Active Comparator): DP-R208 pla+Candesartan 32mg pla+Rosuvastatin 20mg
  Interventions: Drug: Rosuvastatin 20mg; Drug: DP-R208 Placebo; Drug: Candesartan32mg Placebo

INTERVENTIONS:
Drug: DP-R208 — DP-R208 + Candesartan 32mg placebo + Rosuvastatin 20mg placebo
  Arms: CR group
Drug: Candesartan32mg — DP-R208 placebo + Candesartan 32mg + Rosuvastatin 20mg placebo
  Other Names: Candesartan
  Arms: CP group
Drug: Rosuvastatin 20mg — DP-R208 placebo + Candesartan 32mg placebo + Rosuvastatin 20mg
  Other Names: Rosuvastatin
  Arms: PR group
Drug: DP-R208 Placebo — DP-R208 placebo + Candesartan 32mg placebo + Rosuvastatin 20mg
  Arms: CP group; PR group
Drug: Candesartan32mg Placebo — DP-R208 placebo + Candesartan 32mg placebo + Rosuvastatin 20mg
  Arms: CR group; PR group
Drug: Rosuvastatin 20mg Placebo — DP-R208 placebo + Candesartan 32mg + Rosuvastatin 20mg placebo
  Arms: CP group; CR group

SUMMARY:
The purpose of this study is to determine superiority of DP-R208 compare to each monotherapy in patient with hypertension and primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Both man and woman who is over 19years old.
* Hypertension with primary cholesterolemia and satisfy the lab results that Mean msSBP is under 180mmHg and Mean msDBP is under 110mmHg and LDL-C is 250mg/DL or under and Triglycerides is under 400mg/dL

Exclusion Criteria:

* Therapeutic lifestylechange is not enought during the study period
* SBP difference is bigger than 20mmHg or DBP difference is bigger than 10mmHg at screening visit

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mean change of mean seated Systolic Blood Pressure and Percent change of LDL cholesterol | 8weeks

CONTACTS AND LOCATIONS:
Overall Officials: Changkyu Park, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho KI, Kim BH, Park YH, Ahn JC, Kim SH, Chung WJ, Kim W, Sohn IS, Shin JH, Kim YJ, Chang K, Yu CW, Ahn SH, Kim SY, Ryu JK, Lee JY, Hong BK, Hong TJ, Gyu Park C. Efficacy and Safety of a Fixed-Dose Combination of Candesartan and Rosuvastatin on Blood Pressure and Cholesterol in Patients With Hypertension and Hypercholesterolemia: A Multicenter, Randomized, Double-Blind, Parallel Phase III Clinical Study. Clin Ther. 2019 Aug;41(8):1508-1521. doi: 10.1016/j.clinthera.2019.05.007. Epub 2019 Jul 12. PMID 31307833